CLINICAL TRIAL: NCT03878368
Title: A Dietary Intervention Trial to Examine the Effect of Broccoli Bioactives (Specifically Sulforaphane) on Osteoarthritis (OA)
Brief Title: Broccoli In Osteoarthritis
Acronym: BRIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BRIO Protocol V4.0
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2021-10

CONDITIONS: Osteoarthritis
Keywords: Sulforaphane
MeSH Terms: conditions — Osteoarthritis | interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 32 participants with moderate osteoarthritis will eat soup with the active ingredient once-a-day for 4 days-a-week for 3 months.
  Interventions: Dietary Supplement: Sulforaphane
- Control (Active Comparator): 32 participants with moderate osteoarthritis will eat soup without the active ingredient once-a-day for 4 days-a-week for 3 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Sulforaphane — Intervention soup with dietary sulforaphane
  Arms: Intervention
Dietary Supplement: Placebo — Control soup without dietary sulforaphane
  Arms: Control

SUMMARY:
To determine whether dietary sulforaphane (SFN), naturally available from eating broccoli, improves pain in people with knee osteoarthritis (OA), the trial will compare broccoli soup (rich in SFN) with a soup, which does not contain broccoli (control), but looks and tastes the same. Sixty-four participants with moderate osteoarthritis, chosen at random, will either have the broccoli or the control soup. The participants will eat the soup once-a-day, for 4 days-a-week for 3 months.

DETAILED DESCRIPTION:
This is the first clinical trial to test the benefits of eating broccoli on pain and physical function in knee osteoarthritis (OA).

Many fruits and vegetables in the normal human diet contain substances that may improve human health or disease. There is increasingly strong laboratory data that indicate that exposure to these substances at the levels found in the diet influence the way in which osteoarthritis develops. Sulforaphane (SFN) is a naturally occurring substance found in vegetables such as broccoli and is known to have helpful effects on cartilage cells. Sulforaphane derived from broccoli, has a potential role in limiting pain and cartilage destruction in OA.

The investigators have shown that:

* SFN can stop inflammation in mice with OA
* SFN blocks the production of the enzymes which break down cartilage in OA, both in cell cultures and in pieces of cartilage
* SFN enters the joint in participants provided with a high broccoli diet ahead of a knee replacement and alters the types of proteins present in the joint fluid

The investigators aim to discover for the first time in man, whether a broccoli-rich diet will improve pain and physical function in participants with knee osteoarthritis. The study will provide the much-needed preliminary data that will allow the investigators to design a clinical trial to prove that broccoli can be recommended as a helpful food for people with OA.

The trial will compare broccoli soup (rich in SFN) with a soup, which does not contain broccoli (control), but looks and tastes the same. Sixty-four participants with moderate osteoarthritis will either have the broccoli or the control soup, chosen at random. The participants will eat the soup once-a-day, for 4 days-a-week for 3 months. The investigators will measure pain and physical function at the start of the trial, at 6 weeks and at 12 weeks and look at the changes in these. The investigators will also take blood samples and collect urine to measure SFN levels.

ELIGIBILITY:
Inclusion Criteria:

1. Current knee pain, defined as pain in either knee, in the (one) month before Visit 1, for which the patient gives a severity score of at least 4 on a 0-10 numeric rating scale (NRS).
2. The target knee should fulfil the criteria of the American College of Rheumatology (ACR) for knee osteoarthritis defined as knee pain for most days of the prior month and at least one of the following three factors: age over 50 years; morning stiffness of less than 30 minutes; knee crepitus on motion.
3. Kellgren Lawrence grade 2-3
4. Stable analgesic usage (if using) for 4 weeks prior to trial entry and throughout the trial duration
5. Able to adhere to the study visit schedule and other protocol requirements (willing to consume soup intervention).
6. Willing to provide 24 hour urine collection samples (x3)
7. Capable of giving informed consent and the consent must be obtained prior to any screening procedures.

Exclusion Criteria:

1. The presence of any inflammatory arthritis (e.g. gout, reactive arthritis, rheumatoid arthritis, psoriatic arthritis, seronegative spondylarthropathy) or fibromyalgia or metabolic bone disease.
2. Any clinically significant uncontrolled concurrent illness, which, in the opinion of the Investigator, would impair ability to give informed consent or take part in or complete this clinical study.
3. Known or suspected intolerance or hypersensitivity to the investigational product (broccoli) or standardised meal (see section 9.2), closely related compounds, or any of the stated ingredients.
4. Use of an investigational product within 30 days prior to 'run in' period or active enrolment in another drug or vaccine clinical study.
5. Significant knee injury or any knee surgery within the 6 months preceding enrolment in the study.
6. A history of partial or complete joint replacement surgery in the signal knee at any time, listed for knee surgery, or anticipating knee surgery during the study period.
7. Poor tolerability of venepuncture or lack of adequate venous access for required blood sampling during the study period
8. Nutritional deficiency
9. Use of anticoagulant medication (see notes for inclusion exclusion criteria)
10. Use of intra-articular hyaluronic acid in the signal knee within the 3 months preceding enrolment in the study.
11. Use of intra-articular, intra-muscular or oral corticosteroids in the 2 months preceding enrolment.
12. Commencement of non-pharmacological interventions within two months preceding enrolment.
13. Persons less than 50 years
14. Pregnant/lactating women

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
WOMAC (Western Ontario and McMaster Universities Arthritis Index) | Baseline and 12 weeks.
  Change in the WOMAC (Western Ontario and McMaster Universities Arthritis Index) pain subscale.

SECONDARY OUTCOMES:
WOMAC (Western Ontario and McMaster Universities Arthritis Index): Pain | 6 weeks
  Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright
WOMAC (Western Ontario and McMaster Universities Arthritis Index): Physical Function | 6 & 12 weeks
  Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties
WOMAC (Western Ontario and McMaster Universities Arthritis Index): Stiffness | 6 & 12 weeks
  Stiffness (2 items): after first waking and later in the day
11 Point Pain Numerical Rating Scale (NRS): Average overall knee pain severity in the index knee over the past 1 week | 6&12 weeks
  Minimum score '0' to maximum score '10' Lower numerical value is the better outcome
11 Point Pain Numerical Rating Scale (NRS): Worst knee pain severity in the index knee over the past 1 week | 6&12 weeks
  Minimum score '0' to maximum score '10' Lower numerical value is the better outcome
11 Point Pain Numerical Rating Scale (NRS): Global disease activity over the past 1 week | 6&12 weeks
  Minimum score '0' to maximum score '10' Lower numerical value is the better outcome
11 point pain Numerical Rating Scale (NRS): Satisfaction with index knee function over the past 1 week | 6&12 weeks
  Minimum score '0' to maximum score '10' Lower numerical value is the better outcome
11 point pain Numerical Rating Scale (NRS): Average pain in other joints over the past 1 week | 6&12 weeks
  Minimum score '0' to maximum score '10' Lower numerical value is the better outcome
Pain in other joints | 6&12 weeks
  Joint manikin
Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP) | 6&12 weeks
  Self-Assessment
Rescue analgesics/NSAIDs | 6&12 weeks
  Use of rescue analgesics/NSAIDs

CONTACTS AND LOCATIONS:
Overall Officials: Alexander MacGregor, PhD, Study Director — University of East Anglia
Locations (2):
- United Kingdom (2):
  - Norfolk & Norwich University Hospital, Norwich, Norfolk
  - Chapel Allerton Hospital, Leeds, West Yorkshire